CLINICAL TRIAL: NCT01496040
Title: Prospective Monocentric Open Label Non Randomized Uncontrolled Phase I/II Clinical Gene Therapy Protocol for the Treatment of Retinal Dystrophy Caused by Defects in RPE65
Brief Title: Clinical Gene Therapy Protocol for the Treatment of Retinal Dystrophy Caused by Defects in RPE65
Acronym: RPE65
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: BRD 07/08-K; 2011-000418-21 (EudraCT Number)
Record Dates: First submitted 2011-11-24; First posted 2011-12-21 (Estimated); Last update posted 2015-10-07 (Estimated); Status verified 2015-10

CONDITIONS: Leber Congenital Amaurosis
MeSH Terms: conditions — Leber Congenital Amaurosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- rAAV2/4.hRPE65 (Experimental): 3 cohortes of 3 patients each.
  All the patients enrolled in the study will receive a single subretinal injection in one eye. The eye, that will be injected, will be the eye with the poorest visual acuity.
  Interventions: Drug: rAAV2/4.hRPE65

INTERVENTIONS:
Drug: rAAV2/4.hRPE65 — One injection in on eye
  Cohorte 1 : 3 patients will receive one injection of up to 400 microliters of the IMP
  Cohorte 2 : 3 patients will receive one injection of up to 800 microliters of the IMP.
  Cohorte 3 : 3 patients under age of eighteen will receive one injection up to 400 or 800 microliters of the IMP.

SUMMARY:
The purpose of the study is to assess the safety and efficacy of the active substance rAAV-2/4.hRPE65 in patients with Leber Congenital Amaurosis or Congenital severe early-onset retinal degeneration associated with RPE65 mutation.

ELIGIBILITY:
Inclusion Criteria:

* Mutations that code for abnormal RPE65 protein
* Presence of characteristic abnormalities in fundus
* Dramatic reduction of both rods ans cones ERG responses
* Low visual acuity <0.32
* inform consent signed

Exclusion Criteria:

* Patients with chronic conditions such a haematological, cardiac, renal diseases
* Patients with, within the past 6 months, a clinically significant cardiac disease or known congestive heart failure, cardiac rhytm and conduction abnormalities
* Patients with pulmonaty dysfunction
* Patients with suspected rheumatoid arthritis
* Patients with current systemic infection........

Ages: 6 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 9 (Actual)
Dates: Start 2011-09; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
The drug safety evaluation after administration | After administration of the gene therapy product.The patient will be folloed for the duration of the hospital stay, an average of 7 days
  Biodistribution : Urine sampling and nasal secretion will be collected at several time points after administration of the gene therapy product during all the duration of hospital stay, an average of 7 days.

SECONDARY OUTCOMES:
Different efficacy parameters and immune parameters have to be measured to conclude on the overall amelioration of quality of life of enrolled patients | Between Day -120 and Day-7, Day 5, Day 14, Day 30 Day 60, Day 90, Day 120, Day 180, Day 360
  Recording global ERG (electroretinogram)
  Patient efficacy questionnaire
  Testing of far and near visual acuity, color vision, pupillometry, microperimetry and dark adaptation.

CONTACTS AND LOCATIONS:
Overall Officials: Michel WEBER, Professor, Principal Investigator — Nantes University Hospital
Locations (1):
- CHU Nantes, Nantes, France